CLINICAL TRIAL: NCT03646279
Title: Pilot Investigation of a Thoracolumbar Brace for Individuals With Parkinson's Disease
Brief Title: Thoracolumbar Brace for Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Collaborators: AbiliLife (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2015/06/7
Record Dates: First submitted 2018-08-20; First posted 2018-08-24 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single-subject A-B design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Calibrace — The CALIBRACE is a new product designed to improve posture using a front-to-back tensioning system that lifts shoulders up and back.

SUMMARY:
This pilot study looked to see if a new brace would change the way people with Parkinson's Disease positioned their bodies. It also gathered information on the experience of wearing the brace.

ELIGIBILITY:
Inclusion Criteria:

* 50-80 years of age
* Diagnosed with Parkinson's Disease
* Participant self-reports mild difficulty with posture
* Independent in ambulation without an assistive device (i.e., no walker or cane)
* Able to give consent determined via telephone screen assessment or at minimum can follow simple directions
* Able to tolerate 5 minutes of standing or walking at a time per self-report

Exclusion Criteria:

* Rigid or fixed spine, as determined by self-report and use of thoracolumbar flexibility screen
* Symptoms present before the age of 50
* Other neurologic diagnosis, as determined by self-report
* Spinal surgery
* Lives in a nursing home or skilled facility
* Uncorrected vision loss
* Skin that is sensitive to tape or extremely fragile
* Recent surgery (within the last 3 months) that affects mobility, as determined by self-report
* Chest pain at rest or with activity per self report
* Shortness of breath with daily activity per self report
* Severe orthostatic hypotension assessed during in-person screen with sitting and standing blood pressure, evidenced by a 20-point drop in systolic blood pressure or 10-point drop in diastolic blood pressure and symptoms (e.g., dizziness) that don't resolve in 5 minutes.
* High blood pressure 180/110 resting or systolic blood pressure <90 mmHG
* Resting heart rate > 100 bpm or <50 bpm
* Waist circumference < 31" or > 51" that would prevent proper fitting of CALIBRACE.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Postural Alignment - Neck Position | In a single session, 10 data points per phase were collected
  Measured using PostureScreen Mobile Application and all measured bilaterally
  Neck position measured from (EAM to Acrominom)
  * angulation in degrees (flexion values positive/extension values negative)
  * translation in inches (anterior values positive and posterior values negative)
Postural Alignment - Trunk Position | In a single session, 10 data points per phase were collected
  Measured using PostureScreen Mobile Application and all measured bilaterally
  Trunk position measure form Acrominom to Greater Trochanter of femur,
  * angulation in degrees (flexion values positive/extension values negative)
  * translation in inches (anterior values positive and posterior values negative)
Postural Alignment - Hip/Knee Position | In a single session, 10 data points per phase were collected
  Measured using PostureScreen Mobile Application and all measured bilaterally
  Hip/knee position measured from greater trochanter of femur to lateral epicondyle of femur
  * angulation in degrees (flexion values positive/extension values negative)
  * translation in inches (anterior values positive and posterior values negative)

SECONDARY OUTCOMES:
Postural Sway - Center of pressure position | Single session
  The mean center of pressure location measured in root mean squared through the average of three trials of eyes open and the average of three trials of eyes closed.
Postural Sway - Center of pressure velocity | Single session
  The mean center of pressure velocity measured in meters/second through the average of three trials of eyes open and the average of three trials of eyes closed.
Researcher Developed Survey on the Experience of the Brace - No Formal Name or Abbreviation | Single Session
  Survey/interview with seven 4 points Likert-type rating scale (Strongly Disagree, Disagree, Agree, Strongly Agree). High numbers represent more agreement. and three open-ended questions
  There are no total or subscale scores. The frequency of ratings by participants, by the question is what is reported.

IPD SHARING:
Plan to Share IPD: No
This is not currently a plan to share these data with other researchers.